CLINICAL TRIAL: NCT04186403
Title: A Multicenter, Open-label Trial to Evaluate the Safety and Tolerability of Brexpiprazole in the Treatment of Adult Subjects With Borderline Personality Disorder
Brief Title: Evaluating the Safety and Tolerability of Brexpiprazole in the Treatment of Adults With Borderline Personality Disorder (BPD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 331-201-00195; 2019-002897-30 (EudraCT Number)
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prior Brexpiprazole 2-3 Milligrams Per Day (Experimental): Participants who received blinded brexpiprazole 2 to 3 milligrams per day (mg/day) in the previous double-blind trial (NCT04100096), received open-label brexpiprazole 2 to 3 mg/day tablets, orally for up to 12 weeks.
  Interventions: Drug: Brexpiprazole
- Prior Placebo (Experimental): Participants who received blinded brexpiprazole matching placebo in the previous double-blind trial (NCT04100096), received open-label brexpiprazole 2 to 3 mg/day tablets, orally for up to 12 weeks.
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Administered as tablets.
  Other Names: Rexulti; OPC-34712

SUMMARY:
This study evaluates the safety and tolerability of brexpiprazole in the treatment of adults with borderline personality disorder.

ELIGIBILITY:
Inclusion Criteria:

* Participants, who completed the last treatment visit of the previous double-blind brexpiprazole BPD trial and who, in the opinion of the investigator, could potentially benefit from administration of brexpiprazole for the treatment of BPD.
* Male or female outpatients, ages 18 to 65 years, inclusive, at the time of informed consent of the previous double-blind brexpiprazole BPD trial.

Exclusion Criteria:

* Sexually active males or females of childbearing potential (FOCBP) who do not agree to practice 2 different methods of birth control or remain abstinent during the trial and for 30 days after the last dose of IMP. Male participants must also agree not to donate sperm from trial screening/baseline through 30 days after the last dose of investigational medicinal product (IMP).
* Women who are breastfeeding and/or who have a positive pregnancy test result prior to receiving IMP.
* Participants who participated in a clinical trial within 90 days prior to screening/baseline (with the exception of a previous brexpiprazole double-blind BPD trial) or who participated in more than 2 clinical trials within a year prior to screening/baseline.
* Participants who develop a medically significant abnormality.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding sites, contact 844-687-8522, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Rothman B, Brewer C, Chang D, Hobart M, Hefting N, McQuade RD, Grant JE. A randomised study and an extension study of brexpiprazole in patients with borderline personality disorder. Acta Neuropsychiatr. 2024 Nov 19;37:e39. doi: 10.1017/neu.2024.31. PMID 39558901

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 55 investigational sites in Spain, Ukraine, and the United States (US) from 13 January 2020 to 22 September 2021.
Pre-assignment Details: A total of 203 participants with borderline personality disorder (BPD), who completed the previous double-blind trial (NCT04100096) were screened, out of which 201 participants were enrolled in this study. Of the enrolled participants, 90 received 2 to 3 milligrams per day (mg/day) brexpiprazole and 111 received brexpiprazole matching placebo in the previous double-blind trial.
Period: Overall Study
Arm/Group | Prior Brexpiprazole 2-3 Milligrams Per Day | Prior Placebo
Started | 90 | 111
Safety Sample (Safety sample included all participants who received at least 1 dose of investigational medicinal product (IMP).) | 88 | 111
Completed | 71 | 92
Not Completed | 19 | 19
Not completed — Adverse Event | 1 | 8
Not completed — Lost to Follow-up | 7 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 7 | 8
Not completed — Other: Not Related to Covid-19 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled sample included all participants who signed an informed consent form (ICF) and were enrolled into the trial.
Groups:
- Prior Brexpiprazole 2-3 mg/Day: Participants who received blinded brexpiprazole 2 to 3 mg/day in the previous double-blind trial (NCT04100096), received open-label brexpiprazole 2 to 3 mg/day tablets, orally for up to 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Prior Brexpiprazole 2-3 mg/Day | Prior Placebo | Total
Number analyzed (Participants) | 90 | 111 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (10.5) | 32.0 (10.6) | 32.7 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 92 | 163
  Male | 19 | 19 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 72 | 89 | 161
  Race: Black or African American | 7 | 19 | 26
  Race: American Indian or Alaska Native | 2 | 0 | 2
  Race: Asian | 4 | 0 | 4
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Race: Other | 5 | 2 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 15 | 17 | 32
  Ethnicity: Not Hispanic or Latino | 75 | 93 | 168
  Ethnicity: Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and as Per Severity
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial participant administered an IMP and which does not necessarily have a causal relationship with this treatment. TEAEs are defined as AEs with an onset date on or after the start of open-label treatment. The severity of AEs was graded on a 3-point scale: 1=Mild (Discomfort noticed, but no disruption to daily activity), 2=Moderate (Discomfort sufficient to reduce or affect normal daily activity), and 3=Severe (Inability to work or perform normal daily activity).
Time Frame: Signing of ICF up to 30 days post last dose of study drug (up to approximately 16 weeks)
Population: Safety sample included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Brexpiprazole 2-3 mg/Day | Prior Placebo
Number analyzed (Participants) | 88 | 111
Participants
  TEAEs | 30 | 56
  Mild TEAEs | 14 | 37
  Moderate TEAEs | 19 | 30
  Severe TEAEs | 3 | 4

2. Secondary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Potentially clinically significant ECG abnormalities included rate: Bradycardia (vent <=50 beats per minute [bpm] and decrease >=15 bpm); Rhythm: Sinus bradycardia (<=50 bpm and decrease >=15 bpm), absence during baseline and presence of ventricular premature beat post baseline; ST/T morphology: Absence at baseline and presence of symmetrical T-wave inversion post baseline.
Time Frame: Screening up to Week 12
Population: Safety sample included all participants who received at least 1 dose of IMP. 'Number Analyzed' signifies number of participants with available data for the specified measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Brexpiprazole 2-3 mg/Day | Prior Placebo
Number analyzed (Participants) | 88 | 111
Participants
  Bradycardia: number analyzed (Participants) | 75 | 98
  Bradycardia | 0 | 1
  Sinus Bradycardia: number analyzed (Participants) | 75 | 98
  Sinus Bradycardia | 0 | 1
  Ventricular Premature Beat: number analyzed (Participants) | 75 | 99
  Ventricular Premature Beat | 0 | 1
  Symmetrical T-Wave Inversion: number analyzed (Participants) | 75 | 99
  Symmetrical T-Wave Inversion | 0 | 1

3. Secondary Outcome: Number of Participants With Potentially Clinically Significant Vital Sign Abnormalities
Description: Potentially clinically significant vital sign abnormalities included: Heart rate standing in bpm (<50 bpm and decrease >=15 bpm, >120 bpm and increase >=15 bpm); Weight in kilograms (kgs) (decrease >=7%, increase >=7%).
Time Frame: Screening up to Week 12
Population: Safety sample included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Brexpiprazole 2-3 mg/Day | Prior Placebo
Number analyzed (Participants) | 88 | 111
Participants
  Heart Rate Standing | 3 | 1
  Weight Decreased | 7 | 4
  Weight Increased | 9 | 26

4. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities
Description: Potentially clinically significant laboratory abnormalities included serum chemistry: Prolactin >upper limit of normal (ULN) (nanograms per millilitre [ng/ml] in males and females), fasting glucose ≥100 (milligrams per decilitre [mg/dl]), fasting high-density lipoprotein (HDL) cholesterol <40 (men)/ <50 (women) (mg/dl), fasting low-density lipoprotein (LDL) cholesterol ≥160 (mg/dl), fasting cholesterol ≥240 (mg/dl), fasting triglycerides ≥150 (mg/dl); Creatine phosphokinase (CPK)/renal: Creatine kinase >3xULN (units per litre [U/l]), creatinine ≥2.0 (mg/dl), urea nitrogen ≥30 (mg/dl).
Time Frame: Screening up to Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Brexpiprazole 2-3 mg/Day | Prior Placebo
Number analyzed (Participants) | 88 | 111
Participants
  Prolactin (ng/ml)-Males: number analyzed (Participants) | 17 | 17
  Prolactin (ng/ml)-Males | 1 | 0
  Glucose, Fasting (mg/dL): number analyzed (Participants) | 57 | 72
  Glucose, Fasting (mg/dL) | 13 | 11
  HDL Cholesterol, Fasting (mg/dL): number analyzed (Participants) | 54 | 71
  HDL Cholesterol, Fasting (mg/dL) | 22 | 19
  LDL Cholesterol, Fasting (mg/dL): number analyzed (Participants) | 54 | 71
  LDL Cholesterol, Fasting (mg/dL) | 2 | 3
  Cholesterol, Fasting (mg/dL): number analyzed (Participants) | 55 | 72
  Cholesterol, Fasting (mg/dL) | 2 | 7
  Triglycerides, Fasting (mg/dL): number analyzed (Participants) | 54 | 71
  Triglycerides, Fasting (mg/dL) | 13 | 13

5. Secondary Outcome: Change From Baseline in Simpson-Angus Scale (SAS) Total Score
Description: The SAS scale is used to evaluate extrapyramidal symptoms (EPS) and consists of a list of 10 symptoms of Parkinsonism (gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, head rotation, glabella tap, tremor, salivation, and akathisia). Each item is rated on a 5-point scale, with a score range of 0 (absence of symptoms) to 4 (severe condition). The SAS total score is the sum of the scores for all 10 items, possible total score is 0 to 40. Negative change from baseline indicates less symptoms.
Time Frame: Baseline and Week 12
Population: Safety sample included all participants who received at least 1 dose of IMP. Overall number analyzed is the number of participants with data available for analyses. 'Number Analyzed' signifies number of participants with available data for this outcome measure at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Brexpiprazole 2-3 mg/Day | Prior Placebo
Number analyzed (Participants) | 87 | 111
score on a scale
  Baseline | 0.2 (0.9) | 0.1 (0.6)
  Change From Baseline at Week 12: number analyzed (Participants) | 70 | 82
  Change From Baseline at Week 12 | -0.1 (0.7) | 0.0 (0.6)

6. Secondary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Total Score
Description: The AIMS scale consists of 10 items describing symptoms of dyskinesia: Facial and oral movements (items 1-4), extremity movements (items 5 and 6), and trunk movements (item 7), dyskinesias (items 8-10). Each item is rated on a 5-point scale, with a score range of 0 (absence of symptoms) (for item 10, no awareness) to 4 (severe condition) (for item 10, awareness, severe distress). AIMS total score is the sum of the ratings for the first seven items with the possible total scores of 0 to 28. Negative change from baseline indicates less symptoms.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Brexpiprazole 2-3 mg/Day | Prior Placebo
Number analyzed (Participants) | 87 | 111
score on a scale
  Baseline | 0.0 (0.1) | 0.1 (0.8)
  Change From Baseline at Week 12: number analyzed (Participants) | 70 | 83
  Change From Baseline at Week 12 | 0.0 (0.2) | -0.1 (0.9)

7. Secondary Outcome: Change From Baseline in Barnes Akathisia Rating Scale (BARS): Global Clinical Assessment of Akathisia Score
Description: The BARS consists of 4 items related to akathisia: Objective observation of akathisia by the investigator, subjective feelings of restlessness by the participant, subjective distress due to akathisia, and global clinical assessment of akathisia. The fourth item, global clinical evaluation was rated on a 6-point scale, with a score range of 0 (absence of symptoms) to 5 (severe akathisia). Lower scores indicate less symptoms and negative change from baseline indicate less symptoms.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Brexpiprazole 2-3 mg/Day | Prior Placebo
Number analyzed (Participants) | 87 | 111
score on a scale
  Baseline | 0.1 (0.3) | 0.1 (0.3)
  Change From Baseline at Week 12: number analyzed (Participants) | 70 | 83
  Change From Baseline at Week 12 | -0.1 (0.3) | -0.0 (0.5)

8. Secondary Outcome: Number of Participants With Suicidal Ideation and Behavior as Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS was used to assess the suicidality of participants during the study. The assessment included "yes" or "no" responses for 5 questions, each related to suicidal ideation (wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods, active suicidal ideation with some intent, active suicidal ideation with specific plan) and suicidal behavior (preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, suicide). Numeric ratings were provided for suicidal ideation: Score range of 1 (wish to be dead) to 5 (active suicidal ideation with specific plan and intent), higher total scores indicate more suicidal ideation; Suicidal behavior: Score range of 0 (no suicidal behavior) to 4 (actual suicide attempt), higher total scores indicate more suicidal behavior.
Time Frame: Baseline up to Week 12
Population: Safety sample included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Brexpiprazole 2-3 mg/Day | Prior Placebo
Number analyzed (Participants) | 88 | 111
Participants
  Suicidal Ideation | 28 | 28
  Suicidal Behavior | 0 | 2

ADVERSE EVENTS:
Time Frame: Signing of ICF up to 30 days post last dose of study drug (up to approximately 16 weeks)
Description: All-cause mortality: Enrolled sample included all participants who signed an ICF and were enrolled into the trial; Adverse events: Safety sample included all participants who received at least 1 dose of IMP.
Arm/Group | Prior Brexpiprazole 2-3 mg/Day | Prior Placebo
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/111
Serious Adverse Events (participants affected / at risk) | 1/88 | 2/111
Other Adverse Events (participants affected / at risk) | 8/88 | 31/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Brexpiprazole 2-3 mg/Day (N=88) | Prior Placebo (N=111)
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Brexpiprazole 2-3 mg/Day (N=88) | Prior Placebo (N=111)
Fatigue (General disorders) | 1 | 7
Weight increased (Investigations) | 0 | 6
Akathisia (Nervous system disorders) | 1 | 9
Insomnia (Psychiatric disorders) | 5 | 6
Restlessness (Psychiatric disorders) | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT04186403/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT04186403/SAP_001.pdf